CLINICAL TRIAL: NCT02584894
Title: Potentiation of Trauma Exposure in Post-traumatic Stress Disorder by Repeated Transcranial Magnetic Stimulation : A Control Randomized Study
Brief Title: Potentiation of Trauma Exposure in Post-traumatic Stress Disorder by Repeated Transcranial Magnetic Stimulation
Acronym: TETT-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHAO 15- WEH / TETT- STIM
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; trauma exposure; Repeated transcranial magnetic stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Electrocardiography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS 1Hz (Placebo Comparator): Subjects have 8 session of trauma exposure with repeated transcranial magnetic stimulation (rTMS) at 1Hz on dorsolateral prefrontal cortex (1Hz rTMS is describe in the literature to have no effect on the dorsolateral prefrontal cortex). psychoneurological assessment. Electrodermal conductance measure With conductivity meter . Heart rate measure With electrocardiogram
  Interventions: Device: rTMS 1Hz; Behavioral: psychoneurological assessment; Device: conductivity meter; Device: electrocardiogram
- rTMS 10Hz (Experimental): Subjects have 8 session of trauma exposure with repeated transcranial magnetic stimulation (rTMS) at 10Hz on dorsolateral prefrontal cortex (10Hz rTMS is describe in the literature to have effect on the dorsolateral prefrontal cortex). psychoneurological assessment. Electrodermal conductance measure With conductivity meter. Heart rate measure with electrocardiogram
  Interventions: Device: rTMS 10Hz; Behavioral: psychoneurological assessment; Device: conductivity meter; Device: electrocardiogram

INTERVENTIONS:
Device: rTMS 1Hz — trauma exposure + repeated transcranial magnetic stimulation at 1Hz
  Arms: rTMS 1Hz
Device: rTMS 10Hz — trauma exposure + repeated transcranial magnetic stimulation at 10Hz
  Arms: rTMS 10Hz
Behavioral: psychoneurological assessment — psychoneurological assessment
Device: conductivity meter — electrodermal conductance measure
Device: electrocardiogram — heart rate measure

SUMMARY:
The aim of this study is to assess the efficacy in PTSD treatment of concomitant voluntary reactivation of personal traumatic memories with neuromodulation of the right dorsolateral prefrontal cortex using 10Hz rTMS, compared to 1Hz rTMS, during 2 weeks.

DETAILED DESCRIPTION:
Post-Traumatic Stress Disorder (PTSD) is characterized by intrusive and persistent memory of past result from an event causing or able to cause death, be a threat of death, a severe injury or constitute a threat for physical integrity. It is a frequent disorder in general population (8%). In France, The most frequent traumatic events causing PTSD are serious accidents, rape, physical assaults, violence, etc. PTSD treatment involves antidepressant and cognitive and behavioural psychotherapy, which encourage exposure to elements that remind the trauma (memories, circumstances), with the objective of reducing the fear associated with the traumatic memories. Innovative therapeutic strategies aim to improve the psychotherapeutic effect with enhancement drugs or using neuromodulatory techniques, such as repeated transcranial magnetic stimulation (rTMS).

The aim of this study is to assess the efficacy in PTSD treatment of concomitant voluntary reactivation of personal traumatic memories with neuromodulation of the right dorsolateral prefrontal cortex using 10Hz rTMS, compared to 1Hz rTMS, during 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PCLS score >40
* Able to give his written informed consent
* Not participating another study
* Affiliation to a social security system
* Having a PTSD for 3 months
* No treatment modification for 4 weeks (Psychotropic treatment or structured psychotherapy)

Exclusion Criteria:

* Partially deaf with equipment
* people with identified neurological disease
* people with addiction to psychoactive substance
* people who can't conform to tests
* people having a contraindication for rTMS (cochlear implant )
* people suffering from chronicle or acute delusional disorder
* any circumstances making the people unable to understood nature, aim or consequences of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline Score at Clinician administered PTSD scale | inclusion ; 1 months; 3 months
  Score at Clinician administered PTSD scale

SECONDARY OUTCOMES:
Change from baseline Score at PTSD Checklist (self-assessment) | inclusion ; 1 month; 3 months
  Score at PTSD Checklist (self-assessment) for severity of PTSD
Change from baseline Score at PTSD Checklist (self-assessment) for different dimensions of PTSD | inclusion ; 1 month; 3 months
  Score at PTSD Checklist (self-assessment) for severity of different dimensions of PTSD
Change from baseline Score at anxiety and depression item on Hamilton Anxiety Rating Scale (HAM-A) | inclusion ; 1 month; 3 months
  Score at anxiety and depression item on Hamilton Anxiety Rating Scale (HAM-A)
Change from baseline Score at depression item on Hamilton Anxiety Rating Scale (HAM-A) | inclusion ; 1 month; 3 months
  Score at depression item on Hamilton Depression Rating Scale (HAM-D)
Change from baseline heart rate | inclusion ; 1day ; 1 month, 3 months
  heart rate
Change from baseline electrodermal conductance | inclusion ; 1day ; 1 month, 3 months
  electrodermal conductance measure
Adverse effect | inclusion ; 1day ; 1 month, 3 months
  Adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Wissam EL-HAGE, PhD, Principal Investigator — CHRU TOURS

REFERENCES:
- [Background] Quide Y, Witteveen AB, El-Hage W, Veltman DJ, Olff M. Differences between effects of psychological versus pharmacological treatments on functional and morphological brain alterations in anxiety disorders and major depressive disorder: a systematic review. Neurosci Biobehav Rev. 2012 Jan;36(1):626-44. doi: 10.1016/j.neubiorev.2011.09.004. Epub 2011 Sep 24. PMID 21963442
- [Background] Tapia G, Clarys D, Bugaiska A, El-Hage W. Recollection of negative information in posttraumatic stress disorder. J Trauma Stress. 2012 Feb;25(1):120-3. doi: 10.1002/jts.21659. Epub 2012 Jan 25. PMID 22278745
- [Background] Landre L, Destrieux C, Andersson F, Barantin L, Quide Y, Tapia G, Jaafari N, Clarys D, Gaillard P, Isingrini M, El-Hage W. Working memory processing of traumatic material in women with posttraumatic stress disorder. J Psychiatry Neurosci. 2012 Feb;37(2):87-94. doi: 10.1503/jpn.100167. PMID 21971161
- [Background] Landre L, Destrieux C, Baudry M, Barantin L, Cottier JP, Martineau J, Hommet C, Isingrini M, Belzung C, Gaillard P, Camus V, El Hage W. Preserved subcortical volumes and cortical thickness in women with sexual abuse-related PTSD. Psychiatry Res. 2010 Sep 30;183(3):181-6. doi: 10.1016/j.pscychresns.2010.01.015. Epub 2010 Aug 4. PMID 20688488
- [Background] Jaafari N, Rachid F, Rotge JY, Polosan M, El-Hage W, Belin D, Vibert N, Pelissolo A. Safety and efficacy of repetitive transcranial magnetic stimulation in the treatment of obsessive-compulsive disorder: a review. World J Biol Psychiatry. 2012 Mar;13(3):164-77. doi: 10.3109/15622975.2011.575177. Epub 2011 May 30. PMID 21623668